CLINICAL TRIAL: NCT02106273
Title: The Use of LMA-Proseal and Endobronchial Blocker for One Lung Anesthesia, Case Series.
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Prasert Sawasdiwipachai, Instructor, Mahidol University
Other Study IDs: Si154/2011
Record Dates: First submitted 2014-03-30; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Anesthetic Technique; One-lung Ventilation
Keywords: LMA; Bronchial blocker

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bronchial blocker: Pilot study to enroll ASA class I-III patients age between 18-70 years who undergoes thoracic surgery which require one-lung ventilation.
  Interventions: Device: Bronchial blocker (Coopdech, Arndt); Device: LMA-ProsealTM

INTERVENTIONS:
Device: Bronchial blocker (Coopdech, Arndt) — Using bronchial blocker with LMA
  Other Names: Coopdech; Arndt
Device: LMA-ProsealTM

SUMMARY:
An observational pilot study to determine the success rate of using LMA Proseal in conjuction with endobronchial blocker to provide one-lung anesthesia for thoracic surgery.

DETAILED DESCRIPTION:
The use of LMA has gained popularity secondary to benefits confirmed by many literatures. However, LMA is rarely used in thoracic surgery. To enable one-lung ventilation, the LMA need to be used with bronchial blocker. The use of this combination has been reported as a rescue technique in special clinical scenarios, i.e. patient with difficult airway. When used in patient with difficult airway, the LMA will be inserted until proper ventilation achieved, then endobronchial blocker will be subsequently placed through the LMA into the selected main bronchus. The success rate of the the bronchial blocker placement via properly placed LMA has never been studied. This pilot study was designed to evaluate the success rate, the quality of lung collapsed, the dislodgement or other associated problems including some minor complications i.e. postoperative dysphagia, sore throat hoarseness of voice.

ELIGIBILITY:
Inclusion Criteria:

* thoracic surgery that needed one-lung ventilation Exclusion Criteria:patient with
* Restrictive lung disease that needed positive pressure ventilation > 30 cm.H2O
* Mass or hematoma in the mouth which obstruct LMA insertion
* Emergency surgery
* Pregnancy
* Severe infection or active pulmaonary tuberculosis
* Hemoptysis
* Pulmonary nodule > 20 cm. or bronchilal pathology
* Pneumonectomy or sleeve resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA class I-III patients age 18-75 years scheduled for thoracic surgery that required one-lung ventilation
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
success rate | 15 mintues
  can provide one-lung ventilation within 15 mintues

SECONDARY OUTCOMES:
Time consuming in achieving one-lung anesthesia | 15 mintues
  Total time spent to place bronchial blocker into the selected main bronchus shall not exceed 15 minutes. If investigators failed, the study will be terminated and patient will receive appropriate conventional airway management.
Sorethroat | 1 day
  Patient self assessment scale as followed 0 - no sore throat
  1. - mild sore throat (no pain at rest, only with swallowing, does not require intervention)
  2. - moderate sore throat (some discomfort at rest, more with swallowing - but does not need medications)
  3. - severe sore throat (at rest, require analgesics for sore throat)
Hoarseness of voice | 1 day
  Patient assessment scale by visitor as followed 0 - no hoarseness of voice detected, normal voice.
  1. - some hoarseness of voice detected but able to speak in all octaves.
  2. - notable hoarseness of voice, unable to phonate in high pitch.
  3. - marked hoarseness of voice, unable to phonate
Difficulty swallowing | 1 day
  Patient self assessment and visitor assessment in scale as followed. 0 - no problem swallowing. no pain.
  1. - some sore throat (grade 1) with swallowing but able to swallowing both liquid and solid.
  2. - moderate swallowing limitation, only liquid or soft diet swallowing - unable to swallow solid food
  3. - marked swallowing limitation, patient prefers to fast due to pain associated with swallowing. Speech therapist/OT/PT consult to evaluation swallowing problems

CONTACTS AND LOCATIONS:
Overall Officials: Prasert Sawasdiwipachai, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand